CLINICAL TRIAL: NCT02591394
Title: STEPs to Blood Pressure Reduction. A Randomized Clinical Trial of the Stroke Transitions, Education, and Prevention Clinic Versus Usual Care for Post-Stroke Blood Pressure Reduction
Brief Title: STEPs to Blood Pressure Reduction.
Acronym: STEPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding period ended and slow enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Georgetown University (Other)
Responsible Party: Principal Investigator, Anjail Z Sharrief, Assistant Professor of Neurology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-15-0416
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Stroke Prevention; Blood Pressure Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEP Clinic (Experimental)
  Interventions: Behavioral: STEP Clinic
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: STEP Clinic — Patients will visit with STEP clinic staff (including a stroke nurse practitioner or stroke doctor) to receive personalized goals, stroke education (including diet and exercise), instructions to self-monitor using blood pressure cuff, and prescription medications Patient will be scheduled for additional clinic follow-up or be contacted for telephone follow-up for management of your blood pressure. Questionnaires will be administered to determine medication adherence and persistence (following instructions for prescribed medication), disability, depression, cognition, self-efficacy, and sleep apnea. The care plan determined by the STEP clinic will be shared with the patient's primary care provider.
  Arms: STEP Clinic
Behavioral: Usual Care — Patients will complete questionnaires related to medical history and health behaviors prior to initial visit.
  After being seen by the stroke neurologist, patients may be scheduled to return to the stroke clinic according the doctor's recommendations.
  Recommendations for blood pressure and risk factor monitoring will be sent to primary care providers.
  Arms: Usual Care

SUMMARY:
The Stroke Transitions Education and Prevention (STEP) Clinic is a new type of clinic designed for stroke patients and was established to provide a comprehensive approach to stroke risk factor reduction. The goal of this study will be more effective than usual care at reducing blood pressure in patients with poorly controlled blood pressure after an ischemic or hemorrhagic stroke or transient ischemic attack.

DETAILED DESCRIPTION:
STEP clinic patients will receive personalized goals, instructions to self-monitor, a blood pressure monitor, prescription medications, sleep apnea screening, dietary counseling, and more frequent follow-up if needed. A stroke neurologist will see patients in the usual care group and recommendations will be sent to their primary care providers.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18
* Clinical ischemic stroke, intracerebral hemorrhage, or transient ischemic attack
* Plan to discharge home or to short stay inpatient rehab after stroke
* Two of following required:
* History of hypertension (prior to hospitalization)
* Hospital blood pressure ≥ 140/90 on two or more occasions during hospitalization
* Discharge home on blood pressure medication
* Willingness and ability to follow-up in University of Texas Physicians stroke clinic

Exclusion Criteria:

* Modified Rankin scale (mRs) > 3 at enrollment
* Terminal illness
* Chronic kidney disease stage 4 or greater (eGFR < 30)
* Pregnancy
* Symptomatic flow limiting carotid stenosis without plan for intervention prior to clinic visit
* Stroke etiology presumed unrelated to atherosclerotic risk factors (amyloid angiopathy, vasculitis, malignancy associated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-11; Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Daytime ambulatory systolic blood pressure | 6 months

SECONDARY OUTCOMES:
Daytime ambulatory diastolic blood pressure | 6 months
Nighttime ambulatory systolic blood pressure | 6 months
Nighttime ambulatory diastolic c blood pressure | 6 months
Number of patients achieving blood pressure control at 6 months as assessed by ambulatory blood pressure | 6 months
Number of patients achieving blood pressure control at 6 months as assessed by automated office blood pressure | 6 months
Number of participants who are adherent to blood pressure medications | 6 months
Depressive Symptoms as assessed by Patient Health Questionnaire 9 | 6 months
Number of patient monitoring blood pressure at home | 6 months
Satisfaction with Social Roles and activities as measured by NeuroQuality of Life short form | 6 months
Satisfactions with stroke clinic as assessed by Consumer Assessment of Healthcare Providers and Systems Survey | 6 months
Self Efficacy as Assessed by Medication Adherence Self-Efficacy Scale | 6 months
Number of composite cardiovascular events | 6 months
  cardiac death, myocardial infarction, ischemic stroke, hemorrhagic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Anjail Z Sharrief, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Sharrief AZ, Hinojosa E, Cooksey G, Okpala MN, Avritscher EB, Pedroza C, Denny MC, Samuels J, Tyson JE, Savitz SI. Does care in a specialised stroke prevention clinic improve poststroke blood pressure control: a protocol for a randomised comparative effectiveness study. BMJ Open. 2019 Feb 19;9(2):e024695. doi: 10.1136/bmjopen-2018-024695. PMID 30782915